CLINICAL TRIAL: NCT04795102
Title: Effect of "Autogenous Leukocyte Platelet Rich Fibrin- Tooth Graft" Combination Around Immediately Placed Implants in Periodontally Compromized Sites: A Randomized Clinical Trial
Brief Title: Effect of "Autogenous Leukocyte Platelet Rich Fibrin- Tooth Graft" Combination Around Immediately Placed Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalia Rasheed Issa (Other)
Responsible Party: Sponsor-Investigator, Dalia Rasheed Issa, Director, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KD/03/20
Record Dates: First submitted 2021-03-07; First posted 2021-03-12 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Autogenous Tooth Bone Graft; Immediate Implant Placement; L-PRF

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF with ATBG around implant (Experimental): L-PRF clots to cover ATBG around immediately placed dental implants in the extraction sockets
  Interventions: Combination Product: immediate implant placement with ATBG and L-PRF
- ATBG around implant (Active Comparator): ATBG around immediately placed dental implants in the extraction sockets
  Interventions: Combination Product: immediate implant placement with ATBG

INTERVENTIONS:
Combination Product: immediate implant placement with ATBG and L-PRF — immediate implant placement using ATBG as a graft material, with L-PRF
  Arms: L-PRF with ATBG around implant
Combination Product: immediate implant placement with ATBG — immediate implant placement using ATBG as a graft material without L-PRF
  Arms: ATBG around implant

SUMMARY:
Immediate implant placement into fresh extraction sockets is gaining popularity because of fewer clinical procedures and maintenance of bone architecture compared to conventional methods, thus reducing the treatment time and increasing patient satisfaction. In addition, the survival rate of the immediate implantation is comparable to that of the healed implantation sites. Recently, ATBG made from compromised teeth was applied in bone defects and resulted in a good clinical efficacy. Moreover, it is more accepted by patients to use extracted teeth as a bone graft material, especially in the case of immediate implant placement. In 2020, Kizildağ and coworkers studied the outcome of PRF as an adjunct with ATBG on bone healing in rabbit peri-implant osseous defects. They reported that combination of ATBG with PRF contributed to significantly higher new bone formation and better bone/implant contact in rabbits with peri-implant bone defects. The main hypothesis behind this study is that using L-PRF with ATBG following immediate implant placement could promote stabilization of graft particles and enhance new bone formation with a shorter time. Therefore, the purpose of this study was to compare the clinical and radiographic outcomes of ATBG on bone formation with or without L-PRF around immediately placed dental implants in periodontally compromised teeth.

ELIGIBILITY:
Inclusion Criteria:

* Teeth need to be extracted for periodontal reasons with a defect of labial bone (horizontal or vertical bone defect).
* the teeth without acute inflammation.
* no uncontrolled systemic disease which is not suitable for implantation.
* Good systemic and oral health.

Exclusion Criteria:

* patients with systemic diseases or medications known to alter healing processes
* Psychiatric disorders.
* Root canal treated teeth.
* patients undergoing or who had undergone radiation therapy and chemotherapy to the head and neck region during 12 months.
* patients with para-functional habits.
* alcoholics.
* drug abusers.
* heavy smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
clinical evaluation of bone formation around immediately placed dental implants | 9 months
  Changes on bone formation using ATBG with or without L-PRF around immediately placed dental implants in periodontally compromised teeth
radiographic outcome around immediately placed dental implants | 9 months
  the radiographic outcome of ATBG on bone formation with or without L-PRF around immediately placed dental implants in periodontally compromised teeth

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt